CLINICAL TRIAL: NCT02382796
Title: TREATMENT ACCESS PROTOCOL FOR PATIENTS PREVIOUSLY TREATED WITH DACOMITINIB ON A CLINICAL TRIAL IN JAPAN
Brief Title: A Rollover Protocol of Dacomitinib For Patients In Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A7471055
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: NSCLC
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacomitinib (Experimental): 3 dose strengths (45 mg, 30 mg, and 15 mg), continuous oral daily dosing
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Starting at the current dose level in the prior study. Dose reductions and re-escalations are allowed based on tolerability. Patients may continue to be treated with dacomitinib on this protocol as long as there is evidence of clinical benefit in the judgment of the investigator.

SUMMARY:
The purpose of this study to permit continued access to dacomitinib for patients who participated in other dacomitinib monotherapy treatment protocols in Japan and have the potential to derive clinical benefit without unacceptable toxicity from continued dacomitinib treatment.

DETAILED DESCRIPTION:
The intention of the study is to allow continued use of dacomitinib in Japan for patients on closed dacomitinib clinical trials and who continue to experience clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received dacomitinib on another clinical trial in Japan
* Evidence of a personally signed and dated informed consent document

Exclusion Criteria:

* Patients who meet one or more study withdrawal criteria on the prior study
* Participation in other studies involving other investigational drug(s) during study participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Japan (6):
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka City General Hospital Department of Clinical Oncology, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Suntougun, Shizuoka
  - Cancer Institute Hospital,Japanese Foundation for Cancer Research, Koto-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471055&StudyName=Treatment%20Access%20Protocol%20For%20Patients%20Previously%20Treated%20With%20Dacomitinib%20On%20A%20Clinical%20Trial%20In%20Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It is a multi-center,treatment extension study open in Japan only.Eligible participants were those with advanced non-small cell lung cancer who received and tolerated dacomitinib in studies (A7471009 [NCT01360554] and A7471050 [NCT01774721]) in Japan and had the potential to derive continued clinical benefit based on investigator judgment.
Groups:
- Dacomitinib: Participants received continuous daily dosing of dacomitinib at a dose of 45 mg, 30 mg, or 15 mg. The starting dose of dacomitinib on this treatment extension study was the participant's ending dose from the prior studies (A7471009 [NCT01360554] and A7471050 [NCT01774721]). Dacomitinib was provided as tablets for oral administration.
Period: Overall Study
Arm/Group | Dacomitinib
Started | 7
Completed | 0
Not Completed | 7
Not completed — Global deterioration of health status | 1
Not completed — Objective progression or relapse | 3
Not completed — Commercial dacomitinib became available | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received any study medication.
Arm/Group | Dacomitinib
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese): 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Previously Treated With Dacomitinib on the Parent Study in Japan and Who Got Access to Dacomitinib in This Extension Study
Description: To allow access to dacomitinib for participants who received dacomitinib on prior studies (A7471009 [NCT01360554] and A7471050 [NCT01774721]) in Japan and who had the potential to derive continued clinical benefit from single-agent dacomitinib treatment without unacceptable toxicity based upon the investigator's judgment.
Time Frame: 4 years
Population: All participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib
Number analyzed (Participants) | 7
Participants
  7 | 7

2. Secondary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. TEAEs were those with initial onset or increasing in severity on or after the first dose of investigational product administration.
Time Frame: Day1 to up to 28-35 days after last dose, the range of treatment duration was 40-195 weeks
Population: All participants who received any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib
Number analyzed (Participants) | 7
Participants
  AEs: 7 | 7
  SAEs: 7 | 2

ADVERSE EVENTS:
Time Frame: Day1 to up to 28-35 days after last dose, the range of treatment duration was 40-195 weeks
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Dacomitinib
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib (N=7)
Ileus (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib (N=7)
Anaemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Corneal erosion (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Posterior capsule opacification (Eye disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Pleural infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-01-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT02382796/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02382796/SAP_001.pdf